CLINICAL TRIAL: NCT04044248
Title: Single Center Prospective Pilot Study of Combined Transjugular Intrahepatic Portosystemic Shunt Creation Plus Transvenous Obliteration for the Treatment of Gastric Varices
Brief Title: TIPS Plus Transvenous Obliteration for Gastric Varices
Status: Completed | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Ron Gaba, Associate Professor of Radiology & Pathology, University of Illinois at Chicago
Other Study IDs: 2019-0156
Record Dates: First submitted 2019-07-31; First posted 2019-08-05 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Cirrhosis, Liver; Hypertension, Portal; Esophageal and Gastric Varices; Bleeding Gastric; Encephalopathy
Keywords: Liver cirrhosis; Portal hypertension; Gastric varices; Bleeding; Hepatic encephalopathy; Transjugular intrahepatic portosystemic shunt (TIPS); Transvenous obliteration
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal; Esophageal and Gastric Varices; Brain Diseases; Hemorrhage; Hepatic Encephalopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- TIPS-obliteration: Patients undergoing combined transjugular intrahepatic portosystemic shunt (TIPS) creation plus transvenous obliteration for the treatment of gastric varices (GVs).
  Interventions: Device: TIPS-obliteration

INTERVENTIONS:
Device: TIPS-obliteration — Transjugular intrahepatic portosystemic shunt (TIPS) decompression of portal hypertension coupled with transvenous obliteration of gastric varices (GVs).

SUMMARY:
Variceal hemorrhage (VH) from gastric varices (GVs) results in significant morbidity and mortality among patients with liver cirrhosis. In cases of acute bleeding, refractory bleeding, or high risk GVs, the transjugular intrahepatic portosystemic shunt (TIPS) creation and transvenous variceal obliteration procedures have used to treat GVs. While these techniques are effective, each is associated with limitations, including non-trivial rebleeding and hepatic encephalopathy rates for TIPS and aggravation of esophageal varices, development of new or worsening ascites, and formation of difficult to treat ectopic varices for transvenous obliteration. Increasingly, however, TIPS and transvenous obliteration are viewed as complimentary procedures that can be combined to reduce bleeding risk and ameliorate sequelae of portal hypertension. Yet, despite a strong mechanistic basis for their combination, there are few studies investigating the combined effectiveness of TIPS plus transvenous obliteration. Thus, the aim of this single center prospective pilot study is to assess the effectiveness and safety of combined TIPS creation plus transvenous obliteration for the treatment of GVs, with the overall goal of improving the clinical outcomes of patients with VH related to GVs. The work proposed could lead to important advances in the treatment of bleeding complications due to liver cirrhosis.

DETAILED DESCRIPTION:
Liver cirrhosis-or scarring of the liver-occurs with a worldwide prevalence approximating 4.5-9.5%, affecting hundreds of millions of people. Cirrhosis results in 2% of all global mortality, approximating 1 million deaths per year, and affects more than 600,000 persons in the United States. Variceal hemorrhage (VH) from gastroesophageal varices (GEVs) is a leading cause of mortality in patients with liver cirrhosis. Gastric varices (GVs) occur in 5-33% of patients with cirrhotic liver disease and have a bleeding incidence of 25% within 2-years of development, 36% within 3-years, and 44% within 5-years. GVs are associated with high mortality rates approximating 25% at 2-years. First-line therapy in patients who have not bled includes preventative pharmaceuticals, while acute bleeding is typically treated with vasoconstrictive agents and endoscopic variceal ligation or sclerotherapy. In cases of acute hemorrhage, refractory bleeding, or high risk GVs, Interventional Radiology (IR) guided transjugular intrahepatic portosystemic shunt (TIPS) creation is recommended to decompress varices and divert blood flow through a controlled synthetic conduit. In the modern era, TIPS is associated with initial GV bleeding control in greater than 90% of cases. However, GV rebleeding rates after TIPS are non-trivial, widely ranging between 13-53%. Moreover, GVs are widely thought to remain patent and sustain bleeding at low portosystemic pressure gradients (PSGs), as is the case after TIPS. In addition, TIPS can also contribute to high rates hepatic encephalopathy (HE) due to increased portosystemic shunting. Recently, transvenous obliteration techniques-including balloon-occluded retrograde (BRTO) and antegrade (BATO) transvenous obliteration as well as more recent adaptations including coil- (CARTO) and plug-assisted (PARTO) retrograde transvenous obliteration-have been developed with the intent of directly eradicating GVs. While obliteration techniques are associated with high technical success rates approximating 91-100% and low rebleeding incidence less than 5%, the worsened portal hypertension that follows from GV closure results in adverse side effects, including aggravation of esophageal varices (EVs) in 33% of patients, development of new or worsening of ascites in 10% of patients, and formation of difficult to treat ectopic varices.

Traditionally, TIPS and transvenous obliteration have evolved in relative isolation as different philosophical strategies to address VH. TIPS is more commonly utilized in North America and Europe, where portal decompression with or without adjunctive embolization of varices has been a mainstay of endovascular strategy. Conversely, transvenous obliteration evolved in Asia as a direct treatment of VH by obliterating GEVs (particularly GVs) via sclerosis. These approaches were previously viewed as in conflict with one another as obliteration closes GVs but aggravates portal hypertension, whereas TIPS is designed to reduce portal hypertension. Increasingly, however, TIPS and transvenous obliteration are viewed as complimentary procedures that can be combined to reduce bleeding risk and ameliorate sequelae of portal hypertension. Performed together, TIPS and transvenous obliteration result in the elimination of high flow GVs that are at risk for life threatening hemorrhage, with replacement by a man-made endovascular created portosystemic shunt that is not at risk for rupture as well as reduction the risk for post-obliteration EV aggravation, ascites formation, or development of ectopic varices.

Yet, despite a strong mechanistic basis for their combination, there are few studies investigating the effectiveness of combined TIPS plus transvenous obliteration. Thus, the overarching goal of this single center prospective pilot study is to assess the effectiveness and safety of combined TIPS creation plus transvenous obliteration for the treatment of GVs.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Ability to provide written consent
* Endoscopically proven acute or recurrent VH from GVs, or high risk GVs

Exclusion Criteria:

* Prior indwelling TIPS
* Prior endovascular obliteration procedure
* Elevated heart pressures (left or right)
* Heart failure or severe valvular insufficiency
* Severe pulmonary hypertension
* Rapidly progressive liver failure
* Severe or uncontrolled hepatic encephalopathy
* Uncontrolled systemic infection or sepsis
* Unrelieved biliary obstruction
* Polycystic liver disease
* Extensive primary or metastatic hepatic malignancy
* Severe uncontrolled coagulopathy
* Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult persons aged ≥ 18 years with liver disease and endoscopically proven acute or recurrent variceal hemorrhage from gastric varices (GVs) or endoscopically proven high risk GVs referred to Interventional Radiology (IR) for minimally invasive variceal therapy.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Endoscopic gastric varices eradication rate | 6-months
  Effectiveness outcome
Endoscopic esophageal varices aggravation/resolution rate | 6-months
  Effectiveness outcome
Imaging gastric variceseradication rate | 1-year
  Effectiveness outcome
Gastric varices rebleeding rate | 1-year
  Effectiveness outcome
Ascites incidence/improvement rate | 1-year
  Effectiveness outcome

SECONDARY OUTCOMES:
TIPS + transvenous obliteration combined technical success rate | 2-weeks
  Effectiveness outcome
TIPS + transvenous obliteration combined hemodynamic success rate | 2-weeks
  Effectiveness outcome
Procedure related adverse event rate | 30-days
  Safety outcome
Hepatic encephalopathy rate | 1-year
  Safety outcome
Post-TIPS liver failure incidence and degree | 1-year
  Safety outcome
Transplant free survival | 1-year
  Effectiveness outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ron C Gaba, M.D. M.S., Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Saad WE, Wagner CC, Lippert A, Al-Osaimi A, Davies MG, Matsumoto AH, Angle JF, Caldwell S. Protective value of TIPS against the development of hydrothorax/ascites and upper gastrointestinal bleeding after balloon-occluded retrograde transvenous obliteration (BRTO). Am J Gastroenterol. 2013 Oct;108(10):1612-9. doi: 10.1038/ajg.2013.232. Epub 2013 Aug 13. PMID 23939627
- [Result] Gaba RC. Retrograde-Antegrade Accelerated Trap Obliteration: A Modified Approach to Transvenous Eradication of Gastric Varices. J Vasc Interv Radiol. 2017 Feb;28(2):291-294. doi: 10.1016/j.jvir.2016.10.004. PMID 28110759